CLINICAL TRIAL: NCT03672890
Title: Telestroke for Comprehensive Stroke Care in Acute Stroke Ready Hospitals
Acronym: TELECAST
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: NEUR-2017-26226
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Stroke
Keywords: Telestroke; Telemedicine; Stroke; Secondary stroke prevention
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-Telestroke: Retrospective collection of defined metrics for all ischemic stroke patients admitted to the participating ASRH 2 years prior to implementation of an inpatient telestroke service.
- Post-Telestroke: Prospective collection of defined metrics for all ischemic stroke patients admitted to the participating ASRH after implementation of an inpatient telestroke service.
  Interventions: Other: Telestroke

INTERVENTIONS:
Other: Telestroke — Telestroke is an audiovisual communication network that allows for coordination of stroke care from a distant 'hub' site (the telestroke provider location) to an originating 'spoke' site (patient location) in a HIPAA compliant fashion. In TELECAST, inpatient telestroke rounding will be used to oversee the urgent diagnostic stroke evaluation, secondary stroke prevention, health screening & evaluation, and stroke education in patients admitted with stroke.
  Groups: Post-Telestroke

SUMMARY:
TELEstroke for Comprehensive Stroke Care in Acute Stroke Ready HospiTals (TELECAST) is a prospective single-center study evaluating guideline-based acute ischemic stroke care at an Acute Stroke Ready Hospital (ASRH) pre- and post-initiation of a specialist telestroke inpatient rounding service. TELECAST will study the following clinical endpoints: diagnostic stroke evaluation, secondary stroke prevention, health screening and evaluation, stroke education, inpatient complications, and stroke recurrence rates. Additional relevant non-clinical data will include patient and provider satisfaction scores, transfer patterns, and a cost analysis.

DETAILED DESCRIPTION:
Telestroke is a validated intervention that improves the triage and emergent treatment of acute stroke, specifically related to the use of intravenous thrombolysis. Effective urgent stroke evaluation and secondary stroke prevention is also essential to decrease the risk of recurrent stroke, however, there have been no studies to date examining the use of telestroke to improve delivery of non-emergent inpatient stroke care per American Heart Association (AHA) guidelines.

Currently, access to stroke specialist expertise is limited resulting in significant disparities in stroke care. Previous publications have identified that patients in rural areas may receive sub-optimal stroke care that does not follow accepted guideline recommendations. Telestroke is a cost-effective mechanism to deliver specialist stroke care to hospitals that do not have in-person stroke consultation available. The aim of TELECAST is to determine whether specialist telestroke inpatient rounding improves guideline-based acute stroke care when compared to non-specialist stroke care.

The primary outcome of TELECAST is a composite score comprising 4 categories: diagnostic stroke evaluation, secondary stroke prevention, health screening and evaluation, and stroke education. Individual components of the primary outcome were primarily derived from AHA stroke guidelines. Additional outcome measures include individual analyses of the components of the primary outcome as well as the complication rate, stroke recurrence rate, transfer rate, patient and provider satisfaction levels, and a cost-analysis. All outcomes will be assessed at 1 year post-implementation, with data accruement beginning after a 3-month lead in phase.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Patients with the primary diagnosis of ischemic stroke admitted to Fairview Ridges Hospital
* Evidence of stroke on MRI or CT or clinical diagnosis of acute ischemic stroke by the treating stroke service

Exclusion Criteria:

* Patients less than 18 years old
* Patients who leave the hospital against medical advice
* Patients with goals of care that impact the stroke evaluation (i.e. comfort measures)
* Patients who are felt to have an alternative diagnosis
* Patients who are transferred for higher-level stroke care such as endovascular thrombectomy or decompressive craniectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted with a diagnosis of acute ischemic stroke at a participating ASRH two years before and one year after implementation of the telestroke inpatient service.
Sampling Method: Probability Sample
Enrollment: 551 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Composite score of inpatient stroke care (%) | 1 year after implementation of the inpatient telestroke service
  A 23-item global assessment of fundamental inpatient acute ischemic stroke care primarily informed by AHA guidelines/GWTG criteria comprising 4 categories:
  * Diagnostic evaluation (10 items): neurologist evaluation, LDL, HgA1c, troponin, head CT or brain MRI, intracranial vascular imaging, cervical vascular imaging, EKG, telemetry, and outpatient prolonged cardiac monitoring.
  * Secondary prevention (6 items): antiplatelet, anticoagulation, statin, antihypertensives, diabetes management, and carotid revascularization.
  * Health screening & evaluation (4 items): swallow evaluation, cognitive assessment, depression screening, and rehabilitation evaluation.
  * Stroke education (3 items): tobacco cessation counseling, exercise/lifestyle counseling, and signs of stroke.
  An item is not scored when not indicated clinically (for example tobacco cessation in a non-smoker), therefore the composite scores will be reported and analyzed as percentages.

SECONDARY OUTCOMES:
Diagnostic Stroke Evaluation | 1 year after implementation of the inpatient telestroke service
  A 10-item global assessment of inpatient diagnostic stroke evaluation as well as individual analysis of each item.
  Diagnostic evaluation (10 items): neurologist evaluation, LDL, HgA1c, troponin, head CT or brain MRI, intracranial vascular imaging, cervical vascular imaging, EKG, telemetry, and outpatient prolonged cardiac monitoring.
  An item is not scored when not indicated clinically (for example prolonged cardiac monitoring in a patient with known atrial fibrillation), therefore the composite scores will be reported and analyzed as percentages.
Secondary Stroke Prevention | 1 year after implementation of the inpatient telestroke service
  A 6-item global assessment of secondary stroke prevention as well as individual analysis of each item.
  Secondary stroke prevention (6 items): antiplatelet, anticoagulation, statin, antihypertensives, diabetes management, and carotid revascularization.
  An item is not scored when not indicated clinically (for example deferring antiplatelet agents if a patient requires anticoagulation), therefore the composite scores will be reported and analyzed as percentages.
Health Screening & Evaluation | 1 year after implementation of the inpatient telestroke service
  A 4-item global assessment of health screening and evaluation as well as individual analysis of each item.
  Health screening & evaluation (4 items): swallow evaluation, cognitive assessment, depression screening, and rehabilitation evaluation.
  An item is not scored when not indicated clinically, therefore the composite scores will be reported and analyzed as percentages.
Stroke Education | 1 year after implementation of the inpatient telestroke service
  A 3-item global assessment of stroke education as well as individual analysis of each item.
  Stroke education (3 items): tobacco cessation counseling, exercise/lifestyle counseling, and signs of stroke.
  An item is not scored when not indicated clinically (for example tobacco cessation in a non-smoker), therefore the composite scores will be reported and analyzed as percentages.
Composite Stroke Recurrence | Measured at 3 months and at 1 year after discharge
  The composite rate of recurrent TIA, ischemic, or hemorrhagic stroke at 3 months and one year post-stroke admission.

OTHER OUTCOMES:
Acute Stroke Care | 1 year after implementation of the inpatient telestroke service
  Appropriate and timely delivery of acute stroke interventions per AHA guidelines.
Transfer patterns | 1 year after implementation of the inpatient telestroke service
  Transfer rate and discharge destinations. We will also study the impact of changing transfer patterns on baseline patient demographics of the inpatient stroke service at the participating ASRH.
Inpatient complications | 1 year after implementation of the inpatient telestroke service
  Inpatient complications include: hemorrhagic transformation, UTI, PE, pneumonia, DVT, falls, stage II or greater decubitus ulcers, and mortality.
Provider and patient satisfaction | 1 year after implementation of the inpatient telestroke service
  Provider and patient satisfaction with the telestroke service will be assessed with a questionnaire administered to providers and patients receiving the service.
Cost analysis | 1 year after implementation of the inpatient telestroke service
  A cost analysis incorporating the spoke site and the central (hub) site will be performed. Data collected will include hospital cost of admission, hospital admission reimbursement, transfer costs, and operational costs.
Hospital Length of Stay | 1 year after implementation of the inpatient telestroke service
  The number of days of hospitalization for patients admitted with a primary diagnosis of stroke.
Telestroke feasibility | 1 year after implementation of the inpatient telestroke service
  Descriptive data related to the feasibility of telestroke implementation will be collected. This includes time from admission to when the patient is seen, duration of telestroke screen time, and physician, patient, and nursing satisfaction.
14. Composite score of fundamental inpatient stroke care at non-telestroke ASRHs (%), including Fairview Hospitals: Range, Grand Itasca, Lakes, and Northland | 2 years retrospective data and 1 year prospective data after implementation of the inpatient telestroke service at the participating ASRH
  A 23-item assessment of fundamental inpatient stroke care (see primary outcome) at ASRHs within the same stroke network that do not have an inpatient telestroke service. These scores will serve as temporal controls for the primary outcome.
  An item is not scored if it is not indicated clinically (for example tobacco cessation in a non-smoker), therefore the composite scores will be reported and analyzed as percentages.
Composite score of fundamental inpatient stroke care at the CSC hub site (%) | 2 years retrospective data and 1 year prospective data after implementation of the inpatient telestroke service at the participating ASRH
  A 23-item assessment of fundamental inpatient stroke care (see primary outcome) at the CSC hub site. This data will serve to compare the delivery of inpatient stroke care via inpatient telestroke vs. stroke care delivered in person at the hub site.
  An item is not scored if it is not indicated clinically (for example tobacco cessation in a non-smoker), therefore the composite scores will be reported and analyzed as percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Streib, MD, Principal Investigator — University of Minnesota
Locations (5):
- United States (5):
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Grand Itasca Clinic and Hospital, Grand Rapids, Minnesota
  - Fairview Range Medical Center, Hibbing, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jauch EC, Saver JL, Adams HP Jr, Bruno A, Connors JJ, Demaerschalk BM, Khatri P, McMullan PW Jr, Qureshi AI, Rosenfield K, Scott PA, Summers DR, Wang DZ, Wintermark M, Yonas H; American Heart Association Stroke Council; Council on Cardiovascular Nursing; Council on Peripheral Vascular Disease; Council on Clinical Cardiology. Guidelines for the early management of patients with acute ischemic stroke: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Mar;44(3):870-947. doi: 10.1161/STR.0b013e318284056a. Epub 2013 Jan 31. PMID 23370205
- [Background] Powers WJ, Derdeyn CP, Biller J, Coffey CS, Hoh BL, Jauch EC, Johnston KC, Johnston SC, Khalessi AA, Kidwell CS, Meschia JF, Ovbiagele B, Yavagal DR; American Heart Association Stroke Council. 2015 American Heart Association/American Stroke Association Focused Update of the 2013 Guidelines for the Early Management of Patients With Acute Ischemic Stroke Regarding Endovascular Treatment: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2015 Oct;46(10):3020-35. doi: 10.1161/STR.0000000000000074. Epub 2015 Jun 29. PMID 26123479
- [Background] Kernan WN, Ovbiagele B, Black HR, Bravata DM, Chimowitz MI, Ezekowitz MD, Fang MC, Fisher M, Furie KL, Heck DV, Johnston SC, Kasner SE, Kittner SJ, Mitchell PH, Rich MW, Richardson D, Schwamm LH, Wilson JA; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Peripheral Vascular Disease. Guidelines for the prevention of stroke in patients with stroke and transient ischemic attack: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 Jul;45(7):2160-236. doi: 10.1161/STR.0000000000000024. Epub 2014 May 1. PMID 24788967
- [Background] Demaerschalk BM, Berg J, Chong BW, Gross H, Nystrom K, Adeoye O, Schwamm L, Wechsler L, Whitchurch S. American Telemedicine Association: Telestroke Guidelines. Telemed J E Health. 2017 May;23(5):376-389. doi: 10.1089/tmj.2017.0006. Epub 2017 Apr 6. PMID 28384077
- [Background] Alberts MJ, Wechsler LR, Jensen ME, Latchaw RE, Crocco TJ, George MG, Baranski J, Bass RR, Ruff RL, Huang J, Mancini B, Gregory T, Gress D, Emr M, Warren M, Walker MD. Formation and function of acute stroke-ready hospitals within a stroke system of care recommendations from the brain attack coalition. Stroke. 2013 Dec;44(12):3382-93. doi: 10.1161/STROKEAHA.113.002285. Epub 2013 Nov 12. PMID 24222046
- [Background] Wechsler LR, Demaerschalk BM, Schwamm LH, Adeoye OM, Audebert HJ, Fanale CV, Hess DC, Majersik JJ, Nystrom KV, Reeves MJ, Rosamond WD, Switzer JA; American Heart Association Stroke Council; Council on Epidemiology and Prevention; Council on Quality of Care and Outcomes Research. Telemedicine Quality and Outcomes in Stroke: A Scientific Statement for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2017 Jan;48(1):e3-e25. doi: 10.1161/STR.0000000000000114. Epub 2016 Nov 3. PMID 27811332
- [Background] Switzer JA, Demaerschalk BM, Xie J, Fan L, Villa KF, Wu EQ. Cost-effectiveness of hub-and-spoke telestroke networks for the management of acute ischemic stroke from the hospitals' perspectives. Circ Cardiovasc Qual Outcomes. 2013 Jan 1;6(1):18-26. doi: 10.1161/CIRCOUTCOMES.112.967125. Epub 2012 Dec 4. PMID 23212458
- [Background] Meyer BC, Raman R, Hemmen T, Obler R, Zivin JA, Rao R, Thomas RG, Lyden PD. Efficacy of site-independent telemedicine in the STRokE DOC trial: a randomised, blinded, prospective study. Lancet Neurol. 2008 Sep;7(9):787-95. doi: 10.1016/S1474-4422(08)70171-6. PMID 18676180
- [Background] Kepplinger J, Barlinn K, Deckert S, Scheibe M, Bodechtel U, Schmitt J. Safety and efficacy of thrombolysis in telestroke: A systematic review and meta-analysis. Neurology. 2016 Sep 27;87(13):1344-51. doi: 10.1212/WNL.0000000000003148. Epub 2016 Aug 26. PMID 27566746
- [Background] Muller-Barna P, Hubert GJ, Boy S, Bogdahn U, Wiedmann S, Heuschmann PU, Audebert HJ. TeleStroke units serving as a model of care in rural areas: 10-year experience of the TeleMedical project for integrative stroke care. Stroke. 2014 Sep;45(9):2739-44. doi: 10.1161/STROKEAHA.114.006141. PMID 25147327
- [Background] Tarnutzer AA, Lee SH, Robinson KA, Wang Z, Edlow JA, Newman-Toker DE. ED misdiagnosis of cerebrovascular events in the era of modern neuroimaging: A meta-analysis. Neurology. 2017 Apr 11;88(15):1468-1477. doi: 10.1212/WNL.0000000000003814. Epub 2017 Mar 29. PMID 28356464
- [Background] Ovbiagele B, Schwamm LH, Smith EE, Hernandez AF, Olson DM, Pan W, Fonarow GC, Saver JL. Recent nationwide trends in discharge statin treatment of hospitalized patients with stroke. Stroke. 2010 Jul;41(7):1508-13. doi: 10.1161/STROKEAHA.109.573618. Epub 2010 May 27. PMID 20508182
- [Background] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL; American Heart Association Stroke Council. 2018 Guidelines for the Early Management of Patients With Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2018 Mar;49(3):e46-e110. doi: 10.1161/STR.0000000000000158. Epub 2018 Jan 24. PMID 29367334
- [Background] Lavallee PC, Meseguer E, Abboud H, Cabrejo L, Olivot JM, Simon O, Mazighi M, Nifle C, Niclot P, Lapergue B, Klein IF, Brochet E, Steg PG, Leseche G, Labreuche J, Touboul PJ, Amarenco P. A transient ischaemic attack clinic with round-the-clock access (SOS-TIA): feasibility and effects. Lancet Neurol. 2007 Nov;6(11):953-60. doi: 10.1016/S1474-4422(07)70248-X. PMID 17928270
- [Background] Rothwell PM, Giles MF, Chandratheva A, Marquardt L, Geraghty O, Redgrave JN, Lovelock CE, Binney LE, Bull LM, Cuthbertson FC, Welch SJ, Bosch S, Alexander FC, Silver LE, Gutnikov SA, Mehta Z; Early use of Existing Preventive Strategies for Stroke (EXPRESS) study. Effect of urgent treatment of transient ischaemic attack and minor stroke on early recurrent stroke (EXPRESS study): a prospective population-based sequential comparison. Lancet. 2007 Oct 20;370(9596):1432-42. doi: 10.1016/S0140-6736(07)61448-2. PMID 17928046